CLINICAL TRIAL: NCT06304532
Title: Clinical Efficacy Assessment of Alsareen Capsule for the Management of Helicobacter Pylori (H. Pylori) Infection
Brief Title: Clinical Efficacy and Safety Assessment of Alsareen Capsule for the Management of H. Pylori Infection
Status: Completed | Type: Observational
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, Anees ur Rehman, Principal Investigator, Hamdard University
Other Study IDs: HU123
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Helicobacter pylori infection is a major cause of morbidity and mortality worldwide. More than 50% of the global population is estimated to be infected. In 2015, there were approximately 4.4 billion individuals with H pylori infection worldwide. In Pakistan the prevalence of H. pylori infection, highest (63%) in middle age (41-60 years) group while lowest (33%) in teens and pre-teens (<20 years) group. In young age (20-40) and old age (>60 years) groups, the prevalence of H. pylori was 55% and 60% respectively.

In conventional system of medicine H. pylori infection is treated by triple regimen antibiotic therapy that are amoxicillin, clarithromycin and metronidazole along with acid reducing proton pump inhibitor. Due to recurrence of infection this therapy is repeated multiple times resulting in drug resistance and long term side effects. These side effects & a long term impact of H. pylori in patient general health necessitates development of a safe and long term effective therapy.

DETAILED DESCRIPTION:
Introduction:

Peptic ulcers are open sores that develop on the inside lining of stomach and the upper portion of small intestine. The most common symptom of a peptic ulcer is stomach pain. Peptic ulcers include; Gastric ulcers that occur on the inside of the stomach and Duodenal ulcers that occur on the inside of the upper portion of small intestine (duodenum). The most common cause of peptic ulcers infection is the bacterium Helicobacter pylori (H. pylori). Helicobacter pylori infection is a major cause of morbidity and mortality worldwide. The World Health Organization has declared H. pylori as a Class 1 carcinogen.

In conventional system of medicine H. pylori infection is treated by triple regimen antibiotic therapy that are amoxicillin, clarithromycin and metronidazole along with acid reducing proton pump inhibitor. Due to recurrence of infection this therapy is repeated multiple times resulting in drug resistance and long term side effects. These side effects & a long term impact of H. pylori in patient general health necessitates development of a safe and long term effective therapy.

Alsareen is a DRAP registered product of Hamdard Laboratories (Waqf) Pakistan (HLWP). Alsareen is a time tested formulation developed at Hamdard Research Center and it is being used clinically for more than 15 years. This formulation was shared for broader use at Hamdard Matabs since 1.5 years and found satisfactory. The study will be conducted at Shifa ul Mulk Memorial Hospital Hamdard University, Hamdard Matab Nazimabad and Hamdard Matab Arambagh. The sample size of 50 Subjects suffering from H. pylori Infection will be study and managed by Unani Medicine 'Alsareen'.

Epidemiology:

H. pylori prevalence ranges between 85% and 95% in developing countries and between 30 and 50% in developed countries. After the year 2000, the prevalence of H. pylori became lower than before in European countries. However, in Asia, the prevalence remains the same. More than 50% of the global population is estimated to be infected. In 2015, there were approximately 4.4 billion individuals with H pylori infection worldwide. In Pakistan the prevalence of H. pylori infection, highest (63%) in middle age (41-60 years) group while lowest (33%) in teens and pre-teens (<20 years) group. In young age (20-40) and old age (>60 years) groups, the prevalence of H. pylori was 55% and 60% respectively. Typically, around 90% of infected individuals do not have clinical indications or complications of the illness. However, untreated H. pylori infection can last a lifetime leading to chronic gastritis, which can develop into ulcer and carcinoma. This introduces the need for early diagnosis and proper disease therapy.

Clinical presentation:

The combination of retrosternal pain, weight loss, food intolerance and the absence of halitosis signified a 64% accuracy in predicting H. pylori infection. It is not possible to differentiate between H. pylori-positive and H. pylori-negative functional dyspeptics on the basis of clinical presentation and the number of complaints. However, overall symptom score and severity of several symptoms was significantly higher in the H. pylori-positive group.

Study objective:

To conduct an open randomized, multicenter pilot study for the evaluation of clinical efficacy of Alsareen capsule for the management of H pylori infection.

Null hypothesis (H0) There are no significant effects of Unani Medicine 'Alsareen' in the management of H pylori infection.

Alternate hypothesis (H1) Unani medicine 'Alsareen' is clinically effective for the Management of H pylori Infection.

Study Design:

Open label, single arm pilot study. Duration of treatment: 6 weeks of treatment followed by 2 weeks of washing period.

Subjects with clinical presentation of H pylori infection.

Labs Investigations:

Screening Marker:

Blood Anti H pylori

Diagnostic Marker:

Stool Ag for H pylori

Safety Profile:

CBC & ESR LFTs Serum Urea Serum Creatinine These tests will be done in the pathological laboratory of Dow Lab. The subjects meeting the eligibility criteria will be enrolled after taking written informed consent for the study trial. Unani medicine Alsareen will be prescribed to the subjects meeting the selection criteria. The follow ups will be after every two weeks till the end of treatment followed by two weeks washing period.

Subject selection Inclusion criteria Subjects suffering from H. pylori Infection. Subjects having positive test for stool Ag of H. pylori. Subjects over 15 years of age. Subjects agree to use Test Drug throughout the study. Subjects of both sexes are involved. Non pregnant & Non lactating mother. Exclusion criteria Subjects suffering from chronic liver diseases and kidney failure. Subjects currently taking any antibiotics. Subjects suffering from any type of cancer and any other comorbid condition. Subjects having history of adverse drug reaction.

Study Centers:

This study will be conducted in these clinical settings;

1. Shifa ul Mulk Memorial Hospital Hamdard University

Sample Size:

n= 50 subjects.

Study Medicine Details:

Description:

Alsareen is a DRAP registered product of Hamdard Laboratories (Waqf) Pakistan (HLWP) whose ingredients are:

1. Pistacia lentiscus
2. Carum carvi
3. Curcuma caesia

Dosage & Treatment Regimen:

Study medicine dose is 450mg capsule twice daily. Orally before meal with plain water.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from H. pylori Infection.
* Subjects having positive test for stool Ag of H. pylori.
* Subjects over 15 years of age.
* Subjects agree to use Test Drug throughout the study.
* Subjects of both sexes are involved.

Exclusion Criteria:

* Subjects suffering from chronic liver diseases and kidney failure.
* Subjects currently taking any antibiotics.
* Subjects suffering from any type of cancer and any other comorbid condition.
* Subjects having history of adverse drug reaction.
* Pregnant & lactating mother.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consisted of individuals residing in Karachi, specifically focusing on those living near Hamdard University,Gadap Town, a peri-urban area known for its diverse socio-economic and demographic profile. Participants were selected from various neighborhoods to ensure representation across different socio-economic strata.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
H. pylori stool for antigen test will screened before and after treatment. | 42 days
  after administering medication, the H. pylori stool antigen test yielded a negative result, indicating the absence of H. pylori antigens in the stool sample.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Zahoor Zaidi, Principal Investigator — Hamdard University
Locations (1):
- Shifa Ul Memorial Hospital-Hamdard University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No